CLINICAL TRIAL: NCT01363713
Title: A Long-term Open-label Study of DE-114 Ophthalmic Solution in Patients With Allergic Conjunctivitis - Phase 3 -
Brief Title: A Long-term Study of DE-114 Ophthalmic Solution in Patients With Allergic Conjunctivitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Santen Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 01141102
Record Dates: First submitted 2011-05-30; First posted 2011-06-01 (Estimated); Results first posted 2014-09-23 (Estimated); Last update posted 2014-10-06 (Estimated); Status verified 2014-09

CONDITIONS: Allergic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: DE-114 ophthalmic solution

INTERVENTIONS:
Drug: DE-114 ophthalmic solution

SUMMARY:
Safety and efficacy of DE-114 ophthalmic solution will be evaluated in patients with allergic conjunctivitis, in an open-label, multicenter study.

ELIGIBILITY:
Inclusion Criteria:

* Provided signed, written informed consent.
* Has a positive result from a Type I allergy test.
* If a subject is a female of childbearing potential, she must utilize reliable contraceptive throughout the study, and must have a negative urine pregnancy test prior to enrollment into this study.

Exclusion Criteria:

* Females who are pregnant, nursing or planning a pregnancy, or females of childbearing potential who are not using a reliable method of contraception.
* Presence of any abnormality or significant illness that could be expected to interfere with the study.

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Primary Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Santen study sites, Osaka, Japan

RESULTS

PARTICIPANT FLOW:
Groups:
- DE-114 Ophthalmic Solution: DE-114 ophthalmic solution. One drop at a time, 4 times-daily dosing, bilateral topical instillation. A single arm study.
Period: Overall Study
Arm/Group | DE-114 Ophthalmic Solution
Started | 130 (Assessed for eligibility)
ALLOCATED | 130
Completed | 124 (Analysed (n=130))
Not Completed | 6
Not completed — Adverse Event | 1
Not completed — Protocol Violation | 3
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | DE-114 Ophthalmic Solution
Number analyzed (Participants) | 130
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.2 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69
  Male | 61

OUTCOME MEASURES:

1. Primary Outcome: Change in Ocular Itching Score by Visit
Description: Change from baseline in the average of Ocular itching score over the past 3 days. Ocular itching was assessed by the subject and graded on a 5 points scale of 0-4 (0=no itching, 4=incapacitating itch).
  The main purpose of this study is not to confirm but to evaluate safety of long term use of this drug, so primary variable was not defined.
Time Frame: From baseline to 8-week
Measure: Mean (Standard Error); unit: score
Arm/Group | DE-114 Ophthalmic Solution
Number analyzed (Participants) | 130
score
  Change in baseline to visit 2 (Day7) | -0.6 (0.1)
  Change in baseline to visit 3 (Day14) | -0.9 (0.1)
  Change in baseline to visit 4 (Day28) | -1.3 (0.1)
  Change in baseline to visit 5 (Day42) | -1.7 (0.1)
  Change in baseline to visit 6 (Day56) | -2.2 (0.1)

2. Other Pre Specified Outcome: Change in Palpebral Hyperemia Score by Visit
Description: Change from baseline of palpebral hyperemia score. Palpebral hyperemia was assessed by the investigator and graded on a 4 points scale of 0-3 (0=none and 3= extremely severe).
  The main purpose of this study is not to confirm but to evaluate safety of long term use of this drug, so primary variable was not defined.
Time Frame: From baseline to 8-week
Measure: Mean (Standard Error); unit: score
Arm/Group | DE-114 Ophthalmic Solution
Number analyzed (Participants) | 130
score
  Change in baseline to visit 2 (Day7) | -0.3 (0.0)
  Change in baseline to visit 3 (Day14) | -0.3 (0.1)
  Change in baseline to visit 4 (Day28) | -0.6 (0.1)
  Change in baseline to visit 5 (Day42) | -0.7 (0.1)
  Change in baseline to visit 6 (Day56) | -1.0 (0.1)

3. Other Pre Specified Outcome: Change in Bulbar Conjunctiva Hyperemia Score by Visit
Description: Change from baseline of bulbar conjunctiva hyperemia score. Bulbar conjunctiva hyperemia was assessed by the investigator and graded on a 4 points scale of 0-3 (0=none and 3= extremely severe).
  The main purpose of this study is not to confirm but to evaluate safety of long term use of this drug, so primary variable was not defined.
Time Frame: From baseline to 8-week
Measure: Mean (Standard Error); unit: score
Arm/Group | DE-114 Ophthalmic Solution
Number analyzed (Participants) | 130
score
  Change in baseline to visit 2 (Day7) | -0.4 (0.1)
  Change in baseline to visit 3 (Day14) | -0.4 (0.1)
  Change in baseline to visit 4 (Day28) | -0.6 (0.1)
  Change in baseline to visit 5 (Day42) | -0.7 (0.1)
  Change in baseline to visit 6 (Day56) | -0.8 (0.1)

ADVERSE EVENTS:
Time Frame: 8-week
Arm/Group | DE-114 Ophthalmic Solution
Serious Adverse Events (participants affected / at risk) | 0/130
Other Adverse Events (participants affected / at risk) | 9/130
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DE-114 Ophthalmic Solution (N=130)
Nasopharyngitis (Infections and infestations) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No